CLINICAL TRIAL: NCT05207423
Title: Patterns of Care and Clinical Outcomes of Patients With Advanced Non-small Cell Lung Cancer (NSCLC) With EGFR Exon 20 Insertion Mutations
Brief Title: A Chart Review Study of Adults With Advanced NSCLC
Acronym: EXTRACT
Status: Completed | Type: Observational
Sponsor: Takeda (Industry)
Responsible Party: Sponsor
Other Study IDs: TAK-788-4002
Record Dates: First submitted 2022-01-12; First posted 2022-01-26 (Actual); Last update posted 2023-02-28 (Actual); Status verified 2023-02

CONDITIONS: Non-small Cell Lung Cancer (NSCLC)
Keywords: Drug Therapy; Retrospective; Chart review; NSCLC; Mobocertinib; EGFR exon 20 NSCLC; Real World
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Participants With Advanced NSCLC With EGFR Exon-20 Mutations: Participants diagnosed with advanced NSCLC with EGFR exon 20 insertions (ex20ins) mutations who were treated according to routine clinical practice will be observed retrospectively up to 6 months or until the end of follow-up.

SUMMARY:
The main aim is to see how treatment patterns and drugs might improve care for adults with advanced or metastatic NSCLC with epidermal growth factor receptor (EGFR) exon-20 driven mutations. Past medical records will be reviewed. No clinic visits or procedures will be required.

DETAILED DESCRIPTION:
This is a retrospective, observational study in participants with advanced NSCLC with EGFR exon-20 driven mutations. This study will look at clinical outcomes, patterns of care and disease management strategies and healthcare resource utilization (HCRU) in a routine clinical practice setting in the real world.

The study will enroll approximately 218 participants. Participants who were treated at the participating sites between 01 January 2017 and 30 November 2021 will be included. The data will be collected retrospectively at the specialized centers from the participants medical records and notes. All the participants will be assigned to a single observational cohort:

• Participants With Advanced NSCLC With EGFR Exon-20 Mutations

This multi-center study will be conducted in Canada, France and Hong Kong. The overall duration of the study will be 6 months.

ELIGIBILITY:
Inclusion Criteria

1. Histologically/cytologically confirmed diagnosis of locally advanced or metastatic (Stage IIb to IV) NSCLC with EGFR ex20ins mutations (based on the evaluation by the treating center) between 01 January 2017 and 30 November 2021.
2. Followed-up at the site between 01 January 2017 and 30 November 2021 for his/her advanced NSCLC, irrespective of their current survival status.

Exclusion Criteria

1. Participants whose investigator has access to fewer than two registered visits for his/her advanced NSCLC between 01 January 2017 and 30 November 2021.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants who were diagnosed with advanced NSCLC with EGFR ex20ins mutations and who were treated at the participating sites will be included until end of follow-up or death, whichever occurs first.
Sampling Method: Non-Probability Sample
Enrollment: 179 (Actual)
Dates: Start 2022-10-03 (Actual); Primary Completion 2023-02-13 (Actual); Study Completion 2023-02-13 (Actual)

PRIMARY OUTCOMES:
Real-world Progression Free Survival (rwPFS) | Up to 6 months
  rwPFS is defined as the time elapsed from the initiation of a new treatment line to real-world progressive disease (rwPD) or death, whichever occurred first. rwPD: unequivocal increase in visible disease/disease burden or presence of new lesions. Participants will be censored at the end of the line of therapy or date of last contact available.
Real-world Overall Response Rate (rwORR) | Up to 6 months
  Overall response rate (ORR) is the percentage of participants on a treatment line who achieve real-world complete response (rwCR) or real-world partial response (rwPR) as best response per treatment line. rwCR: complete resolution of disease; rwPR: partial reduction in size of visible disease in some, or all, areas without any increase in visible disease.
Confirmed Real-world Overall Response Rate (rwCORR) | Up to 6 months
  ORR is the percentage of participants on a treatment line who achieve confirmed rwCR or rwPR as best response per treatment line. Confirmed responses are responses that persist greater than or equal to (>=) 4 weeks after initial response. rwCR: complete resolution of disease; rwPR: partial reduction in size of visible disease in some or all areas without any increase in visible disease.
Real-world Duration of Response (rwDOR) | Up to 6 months
  rwDOR is defined as the time from the date of first rwCR or rwPR after treatment initiation to the date of the first noted occurrence of progressive disease or death. rwCR: complete resolution of disease, rwPR: partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease.
Real-world Disease Control Rate (rwDCR) | Up to 6 months
  rwDCR is defined as the percentage of participants who have a rwCR, rwPR, or real-world stable disease (rwSD) assessment during the course of a line of therapy, among all participants in that cohort. rwCR: complete resolution of disease, rwPR: partial reduction in size of visible disease in some or all areas without any areas of increase in visible disease, rwSD: no change in overall size of visible disease, or mixed response (some lesions increased, some lesions decreased).
Overall Survival (OS) | Up to 6 months
  OS is defined as the time from the date of advanced disease diagnosis until the date of death. Participants for whom a date of death has not been identified, will be censored at the date of last contact available.
Real-world Time to Treatment Discontinuation (rwTTD) | Up to 6 months
  rwTTD is defined as time from treatment initiation to treatment discontinuation for any reason. Treatment discontinuation is defined as the date of the last drug administered during the same treatment line of therapy or death, whichever occurs earlier. Participants are considered to discontinue treatment if they have advanced to a new line of therapy since the last drug administration, have a recorded date of death, or have no visit activity more than 120 days after the last drug administration.

CONTACTS AND LOCATIONS:
Overall Officials: Study Director, Study Director — Takeda
Locations (30):
- Canada (4):
  - William Osler Health System, Brampton, Ontario
  - Grand River Hospital, Kitchener, Ontario
  - Ottawa Hospital Research Institute., Ottawa, Ontario
  - University Health Network Princess Margaret Cancer Research Tower (PMCRT) The MaRS Centre, East Tower, Toronto, Ontario
- France (20):
  - Centre Hospitalier de Saint-Quentin, Saint-Quentin, Aisne
  - Hopital Nord - CHU Marseille, Marseille, Bouches-du-Rhone
  - Centre Francois Baclesse, Caen, Calvados
  - Centre Georges Francois Leclerc, Dijon, Cote-d'Or
  - CHU Brest - Hopital Morvan, Brest, Finistere
  - Institut Bergonie, Bordeaux, Gironde
  - Hopital Larrey, Toulouse, Haute Garonne
  - Centre Hospitalier de la Region d'Annecy, Pringy, Haute Savoie
  - Hopital Albert Calmette - CHU Lille, Lille, Nord
  - Institut Curie - site de Paris, Paris, Paris
  - CHU Clermont-Ferrand, Clermont-Ferrand, Puy De Dome
  - Centre Leon Berard, Lyon, Rhone
  - Hospices Civils de Lyon, Lyon, Rhone
  - CHU Strasbourg - Nouvel Hopital Civil, Strasbourg, Rhone
  - Centre Hospitalier Regional de la Reunion, Saint-Pierre, Seine Saint Denis
  - Hospital Center Henri Duffaut, Avignon, Vaculuse
  - Centre Hospitalier Intercommunal de Creteil, Créteil, Val De Marne
  - CHU Poitiers - Hopital la Miletrie, Poitiers, Vienne
  - Hopital de Versailles, Versailles, Yvelines
  - Hopital Tenon, Paris
- Hong Kong (6):
  - Pamela Youde Nethersole Eastern Hospital, Hong Kong
  - Prince of Wales Hospital, Hong Kong
  - Princess Margaret Hospital, Hong Kong
  - Queen Elizabeth Hospital, Hong Kong
  - Queen Mary Hospital, Hong Kong
  - Tuen Mun Hospital, Hong Kong

IPD SHARING:
Plan to Share IPD: Yes
Takeda provides access to the de-identified individual participant data (IPD) for eligible studies to aid qualified researchers in addressing legitimate scientific objectives (Takeda's data sharing commitment is available on https://clinicaltrials.takeda.com/takedas-commitment?commitment=5). These IPDs will be provided in a secure research environment following approval of a data sharing request, and under the terms of a data sharing agreement.
Supporting Information: Study Protocol, SAP, ICF, CSR
Access Criteria: IPD from eligible studies will be shared with qualified researchers according to the criteria and process described on https://vivli.org/ourmember/takeda/ For approved requests, the researchers will be provided access to anonymized data (to respect patient privacy in line with applicable laws and regulations) and with information necessary to address the research objectives under the terms of a data sharing agreement.
URL: https://vivli.org/ourmember/takeda/

REFERENCES:
- See also: To obtain more information on the study, click here/on this link. — https://clinicaltrials.takeda.com/study-detail/380405177660454c?idFilter=%5B%22TAK-788-4002%22%5D